CLINICAL TRIAL: NCT03285698
Title: A Randomized, Prospective Trial Comparing the Clinical Outcomes for DermACELL® Compared With Integra® Bilayer Wound Matrix
Brief Title: Comparing the Clinical Outcomes of DermACELL® With Integra® Bilayer Wound Matrix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Georgetown University (Other)
Collaborators: LifeNet Health (Industry)
Responsible Party: Principal Investigator, Christopher Attinger, M.D., Chief, Division of Reconstructive Plastic Surgery, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-0061
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Wounds; Chronic Wounds; Nonmalignant Condition
MeSH Terms: conditions — Wounds and Injuries; Precancerous Conditions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Photographs are submitted and evaluated by a blind, independent assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Integra® (Other): Integra® is a bilayer wound matrix made out of bovine tissue.
  Interventions: Device: Integra®
- DermACELL® (Experimental): DermACELL® is a bilayer wound matrix made out of human tissue.
  Interventions: Device: DermACELL®

INTERVENTIONS:
Device: DermACELL® — DermACELL® is a bilayer wound matrix made out of human tissue and is applied to the wound in standard of care fashion.
  Arms: DermACELL®
Device: Integra® — Integra® is a bilayer wound matrix made out of bovine tissue and is applied to the wound in standard of care fashion.
  Arms: Integra®

SUMMARY:
Both DermACELL® and Integra® Bilayer Wound Matrix are indicated for deep soft tissue coverage and serve as a biological matrix for cellular migration. The current thinking about the utility of these products is to apply over the wound surface and wait until the graft is well vascularized (granular bed/neodermis). At that point a split thickness skin graft can be applied over this area to cover and heal the wound. This study will determine whether human allograft or xenograft will create a durable neodermis that is more supportive of accepting of a split thickness skin graft. Patients who do not receive Split thickness skin grafts will be assigned to the second cohort for observation of healing rates.

DETAILED DESCRIPTION:
This is a prospective, randomized, single site, clinical research trial comparing the clinical outcomes of DermACELL® compared with Integra® Bilayer Wound Matrix in dermal regeneration. A total of 100 subjects will be randomized into either the DermACELL® (n=50) or Integra® Bilayer Wound Matrix (n=50) treatment group. An interim analysis will be performed when both groups have enrolled 25 subjects. Subjects will receive either DermACELL® or Integra® Bilayer Wound Matrix in the operating room for coverage of deep soft tissue defects in the lower extremity. Subjects will then be followed in the outpatient clinic. Once the neodermis has been sufficiently generated, a split thickness skin graft (autograft or allograft) will be applied in the operating room. The split thickness skin graft application site will be then followed to observe viability.

ELIGIBILITY:
Inclusion Criteria:

1. male or female 18-90
2. who have a complex soft tissue defect that extends below subcutaneous tissue (exposed fascia, ligament, tendon, muscle, or bone)
3. wounds that are either acute or chronic (nonhealing wounds greater than 4 weeks but not greater than 2 years in duration)
4. wounds not amendable to primary closure as deemed by the surgeon
5. wounds that have been deemed by the surgeon that any residual infection has been or is being treated upon entry into the clinical trial
6. requiring operative application of a dermoconductive agent
7. extremity wounds have adequate perfusion determined by: palpable pedal pulses, dopplerable pulses, ankle brachial index of >0.7, or transcutaneous oximetry of >0.5
8. renally stable (i.e. CR<3.0, BUN>9.0, eGFR >60)
9. is able to comply to clinical trial requirements

Exclusion Criteria:

1. with a contraindication for the application of a xenograft or allograft
2. untreated infection of soft tissue or bone
3. untreated autoimmune connective tissue disorders
4. body mass index of ≥ 50
5. undergoing chemotherapy/radiation therapy
6. malignancy
7. active liver disease (e.g. hepatitis A-G),
8. previous wound care therapy that included any bioengineered alternative tissue or STSG 30 days prior to enrollment
9. pregnancy
10. enrolled in any other interventional clinical research trial
11. unable or unwilling to comply with study requirements

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2014-04-18 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Time the wound bed takes to heal for split thickness skin graft application | 160 days
  Time (days) required for wound bed preparation (granular bed) for the application of a split thickness skin graft (autograft or allograft) after placement of DermACELL® as compared with Integra® Bilayer Wound Matrix.

SECONDARY OUTCOMES:
Percentage of subjects with complete split thickness skin graft take | 30 days
  The percent of subjects with complete split thickness skin graft (autograft or allograft) take utilizing DermACELL® as compared with Integra® Bilayer Wound Matrix 30 days after split thickness skin graft application.

OTHER OUTCOMES:
Percentage of split thickness skin graft take for wound | 30 days
  The percent of split thickness skin graft (autograft or allograft) take for a wound that receives DermACELL® as compared with Integra® Bilayer Wound Matrix 30 days after split thickness skin graft application.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Attinger, MD, Principal Investigator — Georgetown University
Locations (1):
- Medstar Georgetown University Hospital, Washington D.C., District of Columbia, United States